CLINICAL TRIAL: NCT05078775
Title: Prospective, Single Arm Medical Food Study to Evaluate a Standardized Nonessential Amino Acid Restriction (NEAAR) Medical Food for the Dietary Management of Advanced/Metastatic Pancreatic Cancer
Brief Title: Medical Food for the Dietary Management of Advanced/Metastatic Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faeth Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEAAR-001
Record Dates: First submitted 2021-09-01; First posted 2021-10-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Locally Advanced Unresectable Pancreatic Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nonessential Amino Acid Restriction (NEAAR) Medical Food (Experimental): This is a single arm study in which all subjects will receive NEAAR medical food.
  Interventions: Other: NEAAR Medical Food

INTERVENTIONS:
Other: NEAAR Medical Food — Standardized non-essential amino acid restricted medical food.

SUMMARY:
This is a single arm study evaluating the tolerability and markers of pancreatic cancer with a specially designed medical food restricted in specific amino acids for the dietary management of subjects with locally advanced and unresectable or metastatic pancreatic adenocarcinoma. Subjects who are eligible to receive two FDA approved first line drug therapies, gemcitabine and nab-paclitaxel (gem+nabP), routinely prescribed in combination for pancreatic cancer may be included in this study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent form (ICF) by subject.
2. Histologically or cytologically confirmed pancreatic adenocarcinoma.
3. Locally advanced and unresectable or metastatic pancreatic adenocarcinoma.
4. Eligible for standard of care treatment with the gem+nabP regimen.
5. 18 years of age or older.
6. Measurable disease as determined by RECIST 1.1 (at least one measurable lesion must not have been irradiated in the past).
7. ECOG Performance Status of ≤ 1.
8. Adequate organ function during screening evaluation
9. Available pancreatic adenocarcinoma tissue samples from a primary or metastatic site that has been biopsied within the last 12 months and provide consent for them to be obtained and analyzed by the study sponsor to assist in determining final eligibility. A minimum of five (ten preferred) formalin fixed paraffin embedded (FFPE) archival or fresh tumor tissue slides are required.

Key Exclusion Criteria:

1. Any prior neoadjuvant or adjuvant therapy for pancreatic cancer within 6 months of screening.
2. Any prior therapy for metastatic pancreatic cancer or locally advanced and unresectable pancreatic cancer (except for neoadjuvant or adjuvant therapy as noted above in exclusion criteria 1)
3. Known cerebral metastasis.
4. Diagnosis of another malignancy within the past 2 years (excluding a history of carcinoma in situ of the cervix, superficial non-melanoma skin cancer, or superficial bladder cancer that has been adequately treated, or stage 1 prostate cancer that does not require treatment or requires only treatment with luteinizing hormone-releasing hormone agonists or antagonists if initiated at least 30 days prior to beginning the NEAAR medical food).
5. Body mass index (BMI) <18.5 kg/m2 or >40 kg/m2 or serious or refractive cachexia or anorexia that, in the investigator's judgment, prohibits subjects from having energy or appetite sufficient to reliably engage in a strict medical food regimen for an extended time.
6. Presence of any significant comorbidity including clinically significant cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication), myocardial infarction or unstable angina within the 12 months prior to screening, or any major organ failure.
7. Known hypersensitivity, allergy, or religious restrictions regarding pork or pork-derived products; or known allergy to any of the major food allergens as defined by U.S. law (milk, eggs, fish, Crustacean shellfish, tree nuts, peanuts, wheat, soybeans and sesame); or known allergy or hypersensitivity to , gemcitabine or nab-paclitaxel, PERT products (e.g., Pancreaze), or formulary excipients in these products (refer to the FDA-approved package insert).
8. Major surgery or significant traumatic injury within 14 days of planned start of NEAAR medical food or the anticipation of the need for a major surgical procedure during the study.
9. Unwillingness to consume small quantities of meat products and byproducts (e.g., fish sauce, bone marrow, chicken broth).
10. Diagnosed with an eating disorder, irritable bowel syndrome (IBS), Crohn's disease, ulcerative colitis, or gluten-sensitive enteropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Demonstrate tolerability of the NEAAR medical food. | Through study completion (average of 6 months)
  The primary endpoint is the rate of the most common Grade 3 and 4 adverse event (AE) related to the NEAAR medical food.

SECONDARY OUTCOMES:
Overall response rates | Through study completion (average of 6 months)
  Complete response and partial response using RECIST 1.1
Duration of best response | Through study completion (average of 6 months)
Changes in biomarkers | Through study completion (average of 6 months)
  Absolute and relative change from baseline of disease biomarkers
Progression-free survival | Through study completion (average of 6 months)
  Duration from radiographic documentation of disease to radiographic documentation of progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hendifar, MD, Principal Investigator — Cedars-Sinai
Locations (9):
- United States (9):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Oncology Physicians Network, Glendale, California
  - Cedars-Sinai, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Atlantic Health, Morristown, New Jersey
  - xCures - Virtual Site, Raleigh, North Carolina
  - Sarah Cannon, Nashville, Tennessee
  - Baptist Hospitals of Southeast Texas, Beaumont, Texas

IPD SHARING:
Plan to Share IPD: No